CLINICAL TRIAL: NCT05439902
Title: Efficacy of Alpha-blockers (Tamsulosin) in the Treatment of Symptomatic Dysuria in Multiple Sclerosis in Women
Acronym: ALPHA-SEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIMAO/2021-1/EB-01
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis; Dysuria; Lower Urinary Tract Symptoms; Voiding Dysfunction; Urinary Retention
MeSH Terms: conditions — Multiple Sclerosis; Dysuria; Lower Urinary Tract Symptoms; Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: One month of intervention of drug or placebo followed by one month wash-out period and then final one month intervention with the remaining treatment not received in the first cycle.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin (Experimental)
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — One 0.4mg Tamsulosin capsule taken per day for 30 days
  Arms: Tamsulosin
Drug: Placebo — one placebo capsule per day for 30 days. with identical appearance (color and size) to the experimental drug, composed of microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Multiple sclerosis (MS) is the leading non-traumatic cause of severe acquired disability in young people. The disease is defined by relapses, which can affect all neurological functions depending on the location of the new inflammatory lesion(s). The disease can thus manifest itself through bladder and bowel disorders (BWS), which affect approximately 80% of MS patients in all stages. Lower urinary tract dysfunction has a significant negative impact on the quality of life of patients and places a significant burden on the healthcare system in terms of resource allocation. In addition, there is a risk of long-term chronic renal failure, an infectious risk (recurrent cystitis and/or pyelonephritis, sometimes life-threatening) and a lithiasis risk.

The most frequently observed urinary symptoms are: urinary frequency, urgency with or without urinary incontinence, dysuria and chronic retention of urine. These disorders most often combine bladder hyperactivity and dysuria. This dysuria may be responsible for recurrent urinary tract infections, lithiasis, alteration of renal function.

The only therapeutic class currently used to treat dysuria in MS is alpha-blockers. Tamsulosin, alfusozin and doxazosin induce relaxation of the urethral smooth sphincter and prostatic urethral muscle fibers, facilitating the removal of subvesical obstruction and bladder emptying.

The study investigators hypothesize that treatment with tamsulosin 0.4 mg daily in adult MS patients with dysuria will result in symptom improvement as assessed by the International Prostate Symptom Score (IPSS) and Urinary Symptom Profile (USP) scores, a decrease in post-void residual, and an improvement in urine flow and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient with multiple sclerosis (EDSS score < 7.5).
* Moderate to severe dysuria (IPSS score > 7) due to bladder sphincter dyssynergia confirmed by complete urodynamic workup.
* Patient under stable treatment.

Exclusion Criteria:

* The subject is participating in another category 1 interventional study, or a trial involving a non-CE marked or CE marked off-label medical device or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Hypersensitivity to tamsulosin hydrochloride, including angioedema induced by the drug or any of the excipients.
* History of orthostatic hypotension.
* Severe hepatic impairment.
* Concomitant treatment with diclofenac, warfarin, CYP3A4 inhibitors.
* - Patient with complete urinary retention at the time of the pre-inclusion consultation, requiring management by intermittent self-catheterization or, failing that, an indwelling bladder catheter from the outset.
* Major medical or psychiatric illness that, in the opinion of the investigator, would place the subject at risk or could compromise compliance with the study protocol.
* Presence of another neurological pathology (excluding MS).
* Swallowing problems that compromise oral medication.
* Scheduled cataract surgery within 4 months.
* Pregnant, parturient or breastfeeding patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms between groups | Start of first intervention phase (Day 0)
  Measured using the International Prostate Symptom Scale (IPSS), scoring ranging from 0-35
Urinary symptoms between groups | End of first intervention phase (Day 30)
  Measured using the International Prostate Symptom Scale (IPSS), scoring ranging from 0-35
Urinary symptoms between groups | Start of first intervention phase (Day 60)
  Measured using the International Prostate Symptom Scale (IPSS), scoring ranging from 0-35
Urinary symptoms between groups | End of first intervention phase (Day 90)
  Measured using the International Prostate Symptom Scale (IPSS), scoring ranging from 0-35

SECONDARY OUTCOMES:
Urinary symptoms between groups | Start of first intervention phase (Day 0)
  Measured using the Urinary Symptom Profile (USP) questionnaire: score ranging from 0-39
Urinary symptoms between groups | End of first intervention phase (Day 30)
  Measured using the Urinary Symptom Profile (USP) questionnaire: score ranging from 0-39
Urinary symptoms between groups | Start of first intervention phase (Day 60)
  Measured using the Urinary Symptom Profile (USP) questionnaire: score ranging from 0-39
Urinary symptoms between groups | End of first intervention phase (Day 90)
  Measured using the Urinary Symptom Profile (USP) questionnaire: score ranging from 0-39
Post-mictional residue between groups | Start of first intervention phase (Day 0)
  ml, measured with BladderScan
Post-mictional residue between groups | End of first intervention phase (Day 30)
  ml, measured with BladderScan
Post-mictional residue between groups | Start of first intervention phase (Day 60)
  ml, measured with BladderScan
Post-mictional residue between groups | End of first intervention phase (Day 90)
  ml, measured with BladderScan
Maximum urine flow rate between groups | Start of first intervention phase (Day 0)
  ml/s
Maximum urine flow rate between groups | End of first intervention phase (Day 30)
  ml/s
Maximum urine flow rate between groups | Start of first intervention phase (Day 60)
  ml/s
Maximum urine flow rate between groups | End of first intervention phase (Day 90)
  ml/s
Quality of life linked to urinary dysfunction between groups | Start of first intervention phase (Day 0)
  Qualiveen-30 questionnaire; score 0-4
Quality of life linked to urinary dysfunction between groups | End of first intervention phase (Day 30)
  Qualiveen-30 questionnaire; score 0-4
Quality of life linked to urinary dysfunction between groups | Start of first intervention phase (Day 60)
  Qualiveen-30 questionnaire; score 0-4
Quality of life linked to urinary dysfunction between groups | End of first intervention phase (Day 90)
  Qualiveen-30 questionnaire; score 0-4
Quality of life between groups | Start of first intervention phase (Day 0)
  EQ-5D questionnaire; score 0-100
Quality of life between groups | End of first intervention phase (Day 30)
  EQ-5D questionnaire; score 0-100
Quality of life between groups | Start of first intervention phase (Day 60)
  EQ-5D questionnaire; score 0-100
Quality of life between groups | End of first intervention phase (Day 90)
  EQ-5D questionnaire; score 0-100
Fatigue between groups | Start of first intervention phase (Day 0)
  Modified Fatigue Impact Scale; score 0-84
Fatigue between groups | End of first intervention phase (Day 30)
  Modified Fatigue Impact Scale; score 0-84
Fatigue between groups | Start of first intervention phase (Day 60)
  Modified Fatigue Impact Scale; score 0-84
Fatigue between groups | End of first intervention phase (Day 90)
  Modified Fatigue Impact Scale; score 0-84
Drug safety | End of first intervention phase (Day 30)
  Yes/no occurence of the following adverse events: headache, asthenia, gastrointestinal disorders, orthostatic hypotension
Drug safety | End of first intervention phase (Day 90)
  Yes/no occurence of the following adverse events: headache, asthenia, gastrointestinal disorders, orthostatic hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DROUPY, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France